CLINICAL TRIAL: NCT01806701
Title: Biomarkers of Clinical Response to Cognitive Treatment of PTSD in Youth
Brief Title: Brain Response to Treatment for Pediatric PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Amy Sue Garrett, Principle Investigator, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MH097769; K01MH097769 (NIH)
Record Dates: First submitted 2013-02-27; First posted 2013-03-07 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Emotions; Memory Deficits; Post-traumatic Syndrome
Keywords: fMRI; neuroimaging; PTSD; adolescent; trauma; brain
MeSH Terms: conditions — Memory Disorders; Stress Disorders, Post-Traumatic; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Psychotherapy (Experimental): Trauma-focused Cognitive Behavioral Therapy
  Interventions: Behavioral: Trauma-focused cognitive behavioral therapy

INTERVENTIONS:
Behavioral: Trauma-focused cognitive behavioral therapy — the 'gold-standard' behavioral treatment for children/adolescents with posttraumatic stress disorder
  Other Names: TF-CBT

SUMMARY:
This study will examine how brain activation changes as a result of behavioral treatment for posttraumatic stress disorder (PTSD) in adolescents. The investigators will conduct functional magnetic resonance imaging (fMRI) scans before and after the widely-used trauma-focused cognitive behavioral therapy to better understand how the brain recovers from illness. This study will provide much needed information about brain abnormalities in abused youth, and could lead to improvements in behavioral treatments for patients who do not respond to current treatments.

DETAILED DESCRIPTION:
This is a neuroimaging study of changes in brain function associated with trauma-focused cognitive behavioral therapy (TF-CBT)for abused youth suffering from PTSD. By scanning patients before and after treatment, the investigators will identify mediators (potential mechanisms) of recovery from PTSD.

Childhood maltreatment is unfortunately common, and can lead to significant problems in school, emotional difficulties, and physical ailments. Frequently, abused children develop symptoms of posttraumatic stress disorder (PTSD), such as re-experiencing aspects of the trauma, avoiding trauma-related situations, and suffering from chronic hyperarousal. PTSD can inflict significant stress-related damage on the brain at any age, but may be particularly damaging during developmental periods such as adolescence. Therefore, effective treatments for PTSD in youth are critical, and this depends in part on our ability to understand the neural abnormalities underlying pediatric PTSD, and the brain changes accompanying recovery from PTSD.

TF-CBT is the "gold-standard" treatment for this population however, some patients continue to experience symptoms of PTSD following treatment. Examining neural changes associated with successful treatment may suggest adjunctive or additional steps to enhance recovery in non-responders or partly responsive patients.

The investigators will assess brain activation in response to an emotion-related task in 40 adolescents with PTSD before and after a 12 week TF-CBT treatment, conducted at Stanford University. The fidelity of TF-CBT treatment will be assured through ongoing consultation between clinicians and treatment co-creator Judith Cohen, M.D. Neuroimaging analyses will assess patterns of activation associated with response to TF-CBT. Also, the investigators will scan 30 age-matched healthy controls recruited from the same community, to compare with patients to identify abnormalities in brain structure and function in the PTSD group. Controls will be scanned before and after a 12-week interval as well, to allow analyses of test/retest reliability of fMRI measures in this age group.

ELIGIBILITY:
Inclusion Criteria:

* ages 12-17, history of physical or sexual abuse, witnessing violence, or bullying; and English speaking

Exclusion Criteria:

* receiving other psychotherapy currently, taking medications for a psychiatric disorder currently, history of head injury with loss of consciousness longer than 5 minutes; major medical condition such as epilepsy, diabetes, heart disease, or loss of hearing or vision, developmental disorder such as fragile X, autism, or Down's Syndrome, MRI contraindications including metal in the body from an injury or surgery, non-removeable piercings, or braces, Intelligence Quotient (IQ) < 70; schizophrenia, bipolar disorder, current substance abuse.

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 68 (Actual)
Dates: Start 2013-04; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
functional magnetic resonance imaging (brain activation) | change in brain activation after 4 months of treatment (baseline and 4 months)
  We will use functional magnetic resonance imaging to measure changes in brain activation after 4 months of psychotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Amy S Garrett, Ph.D., Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No